CLINICAL TRIAL: NCT04448860
Title: Validation of Standardized Test Protocols to Assess the Impact of Visual Pathologies in Daily Life Activities
Acronym: PROST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: P19-02; 2019-A00483-54 (Other: IDRCB Number)
Record Dates: First submitted 2020-05-19; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-05

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: optimal Simon two-stage design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retinitis Pigmentosa patients (Experimental): Patients with Retinitis Pigmentosa (RP) at different stages of impairment of the visual field, acuity and sensitivity to contrasts 15 patients will be included in phase 1 versus 36 in phase 2 (15 in step 1 and 21 in step 2).
  Interventions: Behavioral: performance of behavioral locomotion tasks phase 1; Behavioral: performance of behavioral locomotion tasks phase 2
- healthy volunteers patients (Other): 36 patients will be included just in phase 2 (15 in step 1 and 21 in step 2).
  Interventions: Behavioral: performance of behavioral locomotion tasks phase 2

INTERVENTIONS:
Behavioral: performance of behavioral locomotion tasks phase 1 — The performance of behavioral locomotion tasks is performed on 4 visits on pilot phase (2 in real condition and 2 in virtual reality in D1 and M1)
  Arms: Retinitis Pigmentosa patients
Behavioral: performance of behavioral locomotion tasks phase 2 — The performance of behavioral locomotion tasks is performed on 6 visits on validation phase (3 in real condition and 2 in virtual reality in D1, M1 and M12)

SUMMARY:
the incidence of the disease of retinal degenerations with loss of photoreceptors (related to old age or genetic) on patients' daily lives, is poorly characterize without standardized means of measurement (usually performed with functional vision or reading tasks).

self-assessment by a quality of life questionnaire correlated with an assessment of emotional state and direct observation of patients during daily life tasks are the two ways used in a scientific framework to collect data on the difficulties encountered by patients in their daily life.

The aim of this project is to determine the behavioral effects of retinitis pigmentosa (RP) by the effects of performance reductions related to adapting to darkness and visual field restriction. Those assessments will be in real conditions but also in virtual reality (VR).

This tool can be used to measure a therapeutic benefit for new treatments (like gene therapy, retinal implants, intra vitreous injections …) for visual loss patients.

DETAILED DESCRIPTION:
This prospective, longitudinal and non-randomized study will be conducted on 2 groups of people: retinitis pigmentosa's patients ( 1st and 2nd phases) and healthy volunteers patients (2nd phase).

The first phase's aim (named pilot phase) is to determine the optimal parameters to achieve the locomotion test. Fifteen RP's eligible patients will be requiring to 4 sessions of 3 hours to perform tests (Two sessions on real conditions and the two others on virtual reality).

The second phase's aim (named validation phase) is to validate tests to assess the impact of peripheral visual impairment on the sensory and motor performance of patients in their daily life. Firstly 15 RP's patients and 15 healthy volunteers will be included in this phase conducted according to a plan of Simon. 21 additional patients will be including on each group in view of the results on the first step in this 2nd phase.

For each patient, the duration of participation will be of 3 months for the first phase and 14 months for the second phase. The study duration is expected to be 50 months.

ELIGIBILITY:
Inclusion Criteria:

* Gender male or female
* Non-syndromic pigmentary retinopathy: diagnosis confirmed by a specialist (RP patients)
* Pigmentary retinopathy with different damage's levels of visual field, acuity and sensitivity to contrasts (RP patients)
* Visual acuity of both corrected eyes (glasses, lenses) greater than or equal to 8/10 (or ≤ 0.1 logMAR) (Healthy volounteers)
* Normal semi-automated kinetic visual field (Healthy volounteers)
* Not participating in any other clinical trial that may interfere with this study
* Sufficient knowledge of the French language to ensure understanding of the tasks to be performed and the instructions received
* Social insurance
* Consent signed after information by the investigator

Exclusion Criteria:

* Pregnant woman
* Inability to give personal consent
* Cataract surgery in the 3 months before inclusion
* Amblyopia
* Inability to comply with the instructions for the study tasks or to complete the study visits
* MMSE score without visual item ≤ 20/25 for RP patients
* MMSE score with visual item ≤ 25/30 for healthy volunteers
* Drug treatment which may cause motor, visual or cognitive disorders (neuroleptics, etc.) or which may interfere with study evaluations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2023-10-04 (Estimated); Study Completion 2023-10-04 (Estimated)

PRIMARY OUTCOMES:
Pilot calibration phase in a real environment. | Month 1
  Defines the optimal parameters of complexity of standardized behavioral tasks thanks to a mobility test in variable light conditions carried out in a real environment.
Pilot calibration phase in a virtual environment. | Month 1
  Defines the optimal parameters of complexity of standardized behavioral tasks thanks to a mobility test in variable light conditions carried out in a virtual environment.
Validation phase on the motor performance | Month 12
  Validation of tests to assess the impact of peripheral visual impairment on the motor performance of patients in their daily life
Validation phase on the sensory performance | Month 12
  Validation of tests to assess the impact of peripheral visual impairment on the sensory performance of patients in their daily life

SECONDARY OUTCOMES:
Validation of a locomotion test in virtual reality | Day 1 - Month 1- Month 12
  It is to validate the construction of the test and to determine its performance in discriminating nature, its reproducibility and its sensitivity to change
Quality of Life Assessment | Day1-Month 1- Month 12
  Analyze the correlation between the results of patients' quality of life and the results of behavioral tests
Measures of the evolution of the postural parameters | Day1 - Month 1 - Month 12
  Evolution of postural's study parameters is performed by an experimental behavioral study, carried out during the same sessions as the main task of locomotion. The participants' postural stability will be correlated with the patient's visual parameters (acuity, visual field).
Analyze the adverse events during the tasks' assessment | through study completion, an average of 1 year
  Analyze the adverse events that will be collected during the performance of this study

CONTACTS AND LOCATIONS:
Overall Officials: Saddek MOHAND-SAID, MD, Principal Investigator — Centre national d'ophtalmologique des 15-20
Locations (1):
- Centre hospitalier national d'ophtalmologique de 15-20, Paris, France